CLINICAL TRIAL: NCT00353353
Title: The Bread Trial: a Demonstration Trial to Show Effects of Fortification of Food With Both Folic Acid and Vitamin B12
Brief Title: The Bread Trial: Effects of Bread Fortified With Folic Acid and Vitamin B12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen Centre for Food Sciences (Other)
Organization: Wageningen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06/02
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2007-07-09 (Estimated); Status verified 2007-07

CONDITIONS: Healthy
Keywords: no specific conditions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: consumption of fortified bread

SUMMARY:
In the Netherlands fortification of food products is not yet mandatory. One of the major arguments of the Dutch Health Council to advise against mandatory fortification is the possibility of masking of a vitamin B12 deficiency. A possible solution to overcome the possibility of masking is: fortification of foods with both folic acid and vitamin B12. In this study we want to assess the effects of this fortification strategy on markers of folate and vitamin B12 status.

DETAILED DESCRIPTION:
During a 12 week period subjects will consume

* bread fortified with folic acid and vitamin B12 or
* placebo bread (not fortified)

Bread consumption has to be at least 3 slices per day, fortification level is 100mcg folic acid and 6mcg vitamin B12 per 3 slices.

We will study the effect of this fortification strategy on markers of folate and vitamin B12 status.

ELIGIBILITY:
Inclusion Criteria:

* age 50-75y

Exclusion Criteria:

* consumption of < 3 slices of bread/day
* use of B-vitamins in the period three months prior to the study
* treatment with B12-injections in the last 5y
* illness or use of medication interfering with folate or vitamin B12 metabolism

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2006-07; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
serum B12 status
serum folate status

SECONDARY OUTCOMES:
erythrocyte folate;
homocysteine;
MMA;
holoTC

CONTACTS AND LOCATIONS:
Overall Officials: Petra Verhoef, PhD, Principal Investigator — Wageningen University; Ingeborg Brouwer, PhD, Principal Investigator — Wageningen University; Martijn Katan, Professor, Principal Investigator — Wageningen University
Locations (1):
- Wageningen University, Wageningen, Netherlands

REFERENCES:
- [Derived] Winkels RM, Brouwer IA, Clarke R, Katan MB, Verhoef P. Bread cofortified with folic acid and vitamin B-12 improves the folate and vitamin B-12 status of healthy older people: a randomized controlled trial. Am J Clin Nutr. 2008 Aug;88(2):348-55. doi: 10.1093/ajcn/88.2.348. PMID 18689370